CLINICAL TRIAL: NCT01104623
Title: Phase 1 Study of Vocal Acoustic Biomarkers in Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: ADHD - Voice Analysis, Vocal Acoustic Biomarkers in Attention Deficit Hyperactivity Disorder
Acronym: ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: MediTECH Electronic GmbH (Unknown); AudioProfiling, Dr. Joerg Langner (Unknown)
Responsible Party: Principal Investigator, Michael Colla, Dr., Charite University, Berlin, Germany
Other Study IDs: AiF KF2247401-AK9-1
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD - Patients: Adults (18-50 years old). All eligible subjects will experience the voice recording procedure followed by the assessment of adult ADHD diagnostics. The diagnostic guidelines for ADHD in adulthood will be accomplished as outlined by expert consensus of the German Society for Psychiatry, Psychotherapy and Neurology, with a semi-structured clinical interview following the DSM-IV-TR criteria and the ADHD-Checklist (ADHD-CL) for DSM-IV (Hesslinger et al., 2002) to assess the severity of ADHD-Symptoms. Childhood ADHD symptoms will be rated retrospectively amongst others by using the short version (WURS-k) of the Wender Utah Rating Scale (Ward et al., 1993), German version (Retz-Junginger et al., 2002). To strengthen the validity of the ADHD diagnosis the reported symptoms were corroborated by second party reports.
- Healthy Controls: Adults(18-50 years old). All eligible subjects will experience the voice recording procedure followed by the ADHD-Checklist (ADHD-CL) for DSM-IV (Hesslinger et al., 2002. To assess the severity of Non-ADHD, the absence of childhood ADHD symptoms will be rated retrospectively amongst others by using the short version (WURS-k) of the Wender Utah Rating Scale (Ward et al., 1993), German version (Retz-Junginger et al., 2002).

SUMMARY:
The purpose of this study is to detect specific vocal acoustic patterns in the voice of attention deficit hyperactivity disorder (ADHD) patients.

DETAILED DESCRIPTION:
This project aims to develop an objective diagnostic instrument for ADHD through an automatic voice-analysis system, which uses as input the natural speech of the participants. The underlying voice-analysis procedure was developed by J. Langner at Humboldt University of Berlin (Langner 2003). It ignores the semantic content of spoken words and extracts prosodic and sound features from the speech.

Aims of the study:

* deliver optimized multivariate logistic regression models of prosodic and sound properties of speech for ADHD.
* observe sensitivity and specificity of the voice-analysis procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50.
2. Written informed consent.
3. Adult ADHD / Non-ADHD according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV)
4. Normal vocal functioning, negative history for voice or laryngeal disorders.
5. Currently euthyroid condition; in case of past history of thyroid disease and need for current pharmacological treatment, patient needs to be on stable medication for at least 4 weeks.

Exclusion Criteria:

1. Exclusion of borderline and antisocial personality disorder, assessed by the German version of the SCID-II (Fydrich et al., 1997).
2. Exclusion of schizophrenia and psychotic disorders not otherwise specified.
3. Exclusion of Epilepsia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: German speaking: Adults, age 18-50 years.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Colla, PhD, Study Chair — Center for ADHD Research, Department of Psychiatry, Charite - University Medicine Berlin
Locations (1):
- Center for ADHD Research, Department of Psychiatry, Charite - University Medicine, Berlin, Germany

REFERENCES:
- [Background] Hamdan AL, Deeb R, Sibai A, Rameh C, Rifai H, Fayyad J. Vocal characteristics in children with attention deficit hyperactivity disorder. J Voice. 2009 Mar;23(2):190-4. doi: 10.1016/j.jvoice.2007.09.004. Epub 2007 Dec 21. PMID 18082369
- [Background] Banse R, Scherer KR. Acoustic profiles in vocal emotion expression. J Pers Soc Psychol. 1996 Mar;70(3):614-36. doi: 10.1037//0022-3514.70.3.614. PMID 8851745
- See also: ADHD - Voice Analysis — http://idw-online.de/pages/de/news345028